CLINICAL TRIAL: NCT01518504
Title: Effects of Thoracic Mobilization on Shoulder Range of Motion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-16286
Record Dates: First submitted 2011-12-01; First posted 2012-01-26 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Shoulder Range of Motion in Healthy Individuals
Keywords: Thoracic; Manipulation; Manual Therapy; Mobilization; Shoulder; Range of Motion
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thoracic Mobilization (Experimental): The subject will be in a prone position and the physical therapist will first identify the upper thoracic spine region. The physical therapist will then cross his or her hands and place them on opposite sides of the spinous processes using the pisiforms as the contact area. The subject will be asked to exhale and upon exhalation the physical therapist will apply a small amplitude, quick thrust at end of range.
  Interventions: Other: Thoracic Mobilization
- Sham (Sham Comparator): The subject will be in a prone position and the physical therapist will first identify the upper thoracic spine region. The physical therapist will then cross his or her hands and place them on opposite sides of the spinous processes using the pisiforms as the contact area. The subject will be asked to exhale and upon exhalation the physical therapist will not apply any other force than light hand contact.
  Interventions: Other: Sham

INTERVENTIONS:
Other: Thoracic Mobilization — The subject will be in a prone position and the physical therapist will first identify the upper thoracic spine region. The physical therapist will then cross his or her hands and place them on opposite sides of the spinous processes using the pisiforms as the contact area. The subject will be asked to exhale and upon exhalation the physical therapist will apply a small amplitude, quick thrust at end of range.
  Other Names: manipulation; Grade V joint mobilization; small amplitude, quick thrust mobilization/manipulation
  Arms: Thoracic Mobilization
Other: Sham — The subject will be in a prone position and the physical therapist will first identify the upper thoracic spine region. The physical therapist will then cross his or her hands and place them on opposite sides of the spinous processes using the pisiforms as the contact area. The subject will be asked to exhale and upon exhalation the physical therapist will not apply any other force than light hand contact.
  Arms: Sham

SUMMARY:
The purpose of this study is to investigate the effect of thoracic spine joint manipulation versus a sham intervention on active and passive shoulder flexion (elevation), external rotation, and internal rotation range of motion.

DETAILED DESCRIPTION:
Many individuals who have a primary complaint of shoulder pain often demonstrate deficits in glenohumeral and scapulothoracic mobility. Typically individuals will have limitations in shoulder range of motion, specifically, flexion (elevation) as well as external and internal rotation. Although the glenohumeral joint is the primary joint for shoulder motion adjacent joints such as the sternoclavicular, acromioclavicular, scapulothoracic, and thoracic spine also contribute to maximal shoulder motion. Limited shoulder motion may be a result of joint hypomobility, muscle inhibition, or pain. Typically interventions such as stretching and joint mobilization/manipulation are directed at the glenohumeral joint to improve shoulder motion, but little is known about interventions targeting adjacent sites which may also improve shoulder range of motion. This study will evaluate the effect of thoracic spine joint manipulation on active and passive shoulder range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Adults 19-45 years

Exclusion Criteria:

* Individuals who are pregnant
* History of cervical or thoracic surgery
* Bone or joint disease
* Current infection or tumor
* Osteopenia/osteoporosis
* Spinal fracture
* Rheumatologic pathologies

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Changes in Shoulder Range of motion | Single Study Visit
  To determine changes in shoulder active and passive range of motion following one of two intervention protocols. Changes will be measured by examining shoulder range of motion in three directions: Shoulder flexion, internal rotation and external rotation.
  We hypothesize that the use of a thoracic spine joint manipulation will increase shoulder range of motion in flexion (elevation) as well as external and internal rotation to a greater degree than a sham mobilization.

CONTACTS AND LOCATIONS:
Overall Officials: Terry L Grindstaff, PHD,PT,ATC, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States